CLINICAL TRIAL: NCT06114888
Title: Optimizing Care for Children Hospitalized With Community-acquired Pneumonia: a Feasibility Randomized Controlled Trial of a Diagnostic Intervention
Brief Title: Optimizing Care for Children Hospitalized With Community-acquired Pneumonia: Novel Diagnostics
Acronym: PRESTO-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jeffrey (Other)
Responsible Party: Sponsor-Investigator, Jeffrey, Associate Professor, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HHS-CB 2023-Pernica-1
Record Dates: First submitted 2023-10-30; First posted 2023-11-02 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Community-acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Intervention Model Description: Participants randomized to usual care or usual care + diagnostic intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MeMed BV (Experimental)
  Interventions: Diagnostic Test: MeMed BV + Usual Care
- Usual Care (Active Comparator)
  Interventions: Other: Usual Care Alone

INTERVENTIONS:
Diagnostic Test: MeMed BV + Usual Care — We will aim to have blood drawn for MeMed BV testing within 24 hours of the first dose of IV antibiotics. We will then aim to have test results back within 24 hours of sampling.
  Arms: MeMed BV
Other: Usual Care Alone — Usual care can involve oxygenation support, ventilatory support, intravenous fluids, and antibiotics, or any combination of these.
  Arms: Usual Care

SUMMARY:
Children are commonly hospitalized because of community-acquired pneumonia. Despite the fact that many of these children have viral disease, a majority is treated with antibiotics. These antibiotics will not accelerate recovery in those with viral pneumonia and can cause harm. We are interested in exploring whether the MeMed BV - a composite biomarker assay - could be used to improve antibiotic prescribing in these children by identifying those who likely have viral disease. This proposal describes a feasibility randomized trial of this diagnostic intervention.

ELIGIBILITY:
Inclusion Criteria:

* children with a history of fever who are hospitalized with CAP (ie. 'severe CAP') as per the clinical team and who have abnormal chest imaging (eg. radiograph, ultrasound) will be eligible. They must also have at least one of the following:

  1. documented tachypnoea (>60 bpm for age <1 y, >50 bpm for 1-2 y, >40 bpm for 2-4 y, and >30 bpm for >4 y);
  2. cough on exam or by history;
  3. increased work of breathing on exam; or
  4. auscultatory findings (eg. focal crackles, bronchial breathing) consistent with CAP.

Exclusion Criteria:

* Children will be excluded from if they have received >48h of intravenous antibiotics (eg. if transferred from another healthcare facility) or if they have a lobar consolidation that occupies the majority of a lobe on imaging, a pleural effusion that occupies more than ¼ of a lung field, or a positive blood culture for a bacterial pathogen (not a contaminant). Examples of CAP pathogens include S. pneumoniae, S. pyogenes (group A streptococcus), S. aureus, S. anginosus. Examples of contaminants that would be ignored include the coagulase-negative staphylococci and Bacillus spp. Children will also be excluded if they have any of the following: chronic lung disease, congenital heart disease (requiring treatment or with exercise restrictions), malignancy, immunodeficiency (primary, acquired, or iatrogenic), a separate episode of pneumonia previously diagnosed within the past 2 weeks, or lung abscess diagnosed within the past six months. Children will not be eligible to participate more than once.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-04-17 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Consent success | Day 0
  The proportion of potentially eligible participants who consent
MeMed BV test timing | before Day 2
  The proportion of participants randomized to the diagnostic intervention who successfully have the MeMed BV performed within 24 h of receipt of the initial dose of IV antibiotics
MeMed BV test result reporting | before Day 3
  The proportion of participants randomized to MeMed BV testing that have a test result available within 48h of sampling
MeMed BV test result initial adherence | before Day 4
  The proportion of participants found to be high risk for viral infection that successfully have their antibiotics stopped within 24 hours of the test result becoming available
MeMed BV test result delayed adherence | before Day 15
  The proportion of participants (who successfully had their antibiotics stopped) that do not have them restarted specifically for CAP treatment prior to discharge
Losses to followup | before Day 30
  The proportion of participants lost to follow-up

SECONDARY OUTCOMES:
Early clinical response | Day 4
  This is defined as:
  i) clinical improvement in fever, work of breathing, oral intake, and activity level, AND ii) lack of receipt of additional antimicrobials beyond those already being given at baseline (for the control group) or as indicated by MeMed BV testing (for those randomized to the intervention group)
Days of antibiotics given specifically for CAP before hospital discharge | Before discharge
Days of antibiotics given specifically for CAP after hospital discharge and before day 30 | after hospital discharge and before day 30
Time to resolution of fever | Before discharge
Time to resolution of difficulty breathing | Before discharge
Time to resolution of hypoxaemia | Before discharge
Length of stay in hospital | Before discharge
Repeat hospitalization for CAP | After discharge and before day 30
Unscheduled ED or urgent care visits | After discharge and before day 30
Unscheduled primary care visits | After discharge and before day 30
Development of complicated pneumonia | Before Day 30
  Complicated defined by effusion, empyaema, necrotizing pneumonia
Acceptability of care plan to caregiver | Baseline
Acceptability of care plan to caregiver | Day 30

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided